CLINICAL TRIAL: NCT04651998
Title: Effect of Carotid Artery Stent on Evoked Cerebral Blood Oxygenation and Neurocognitive Functioning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Collaborators: Minhang Hospital, Fudan University (Unknown); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); RenJi Hospital (Other); ShuGuang Hospital (Other)
Responsible Party: Principal Investigator, Yueqi Zhu, Principal Investigator, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Other Study IDs: CAS-fNIRS
Record Dates: First submitted 2020-11-24; First posted 2020-12-03 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2023-06

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid artery stent, functional near-infrared spectroscopy, vascular cognitive impairment,
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MMSE, MoCA, functional near-infrared spectroscopy — MMSE and MoCA are used for cognitive test before carotid artery stent implant and 6 months later. Cerebral blood oxygenation is evaluated by functional near-infrared spectroscopy under the mental task before and after revascularization within one week, 6 months later respectively.

SUMMARY:
Cerebral hemodynamic compromise from internal carotid artery stenosis may be a cause of vascular cognitive impairment that is amenable to treatment by revascularization. The effect of carotid artery stent on evoked cerebral blood oxygenation and neurocognitive functioning will be evaluated by functional near-infrared spectroscopy. Carotid artery stent could benefit cerebral blood oxygenation after stent and improving neurocognitive functioning after 6 months.

DETAILED DESCRIPTION:
Patients with high grade internal carotid artery stenosis intended to carotid artery stent are brought to this study. Global cognitive function and evoked cerebral blood oxygenation are evaluated before and after stent, followed up at 6 months later. Mini-Mental State Examination(MMSE) and Montreal Cognitive Assessment (MoCA) are used for the global cognitive test. Evoked cerebral blood oxygenation is evaluated using functional near-infrared spectroscopy(fNIRS) through performing mental task( N-back task, Go/no go task, and verbal fluency task ). All the patients from different centers are conducted the test at the only main center by one doctor. The parameter of fNIRS and score of cognitive test of each patient are compared before and after stent.

ELIGIBILITY:
Inclusion Criteria:

1. 35-80 years old
2. Severe carotid stenosis (MRA or CTA confirmed stenosis rate of 70% - 99%, NASCET standard)
3. Asymptomatic or mild stroke (NIHSS ≤ 3) or TIA
4. Agree to participate in the clinical trial and sign the informed consent

Exclusion Criteria:

1. Severe stenosis or occlusion of vertebrobasilar artery and other intracranial arteries (70% - 99%)
2. Left ventricular ejection fraction < 50% or heart failure
3. Other types of dementia have been diagnosed
4. Severe depression, mental illness, epilepsy
5. Not cooperating with cognitive task evaluation

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high grade carotid artery stenosis treated with carotid artery stent from 5 hospitals.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of cognitive function score | MMSE score at baseline, 6 months after revascularization. Change of the score is calculated.
  Mini-mental State Examination (0-30 points), the higher the score, the better the cognitive function

SECONDARY OUTCOMES:
Parameter of evoked cerebral blood oxygenation | Evoked cerebral blood oxygenation evaluated after stent immediately, 6 months later, compared with that at baseline.
  Means of HbO detected by functional near-infrared spectroscopy
Parameter of evoked cerebral blood oxygenation | Evoked cerebral blood oxygenation evaluated after stent immediately, 6 months later, compared with that at baseline.
  Skewness of HbO detected by functional near-infrared spectroscopy
Parameter of evoked cerebral blood oxygenation | Evoked cerebral blood oxygenation evaluated after stent immediately, 6 months later, compared with that at baseline.
  kurtosis of HbO detected by functional near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Yueqi Zhu, PhD, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No